CLINICAL TRIAL: NCT04667091
Title: Comparing the Effects of Positional Release Technique Versus Myofascial Release Technique of Gluteus Medius in the Management of Patellofemoral Pain Syndrome - A Randomized Control Trial
Brief Title: Comparing the Effects of Positional Release Technique Versus Myofascial Release Technique of Gluteus Medius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Priyanka Ratan Kumar, Dr. Priyanka Ratan Kumar (PT), Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-1542
Record Dates: First submitted 2020-12-03; First posted 2020-12-14 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Anterior knee pain; Gluteus medius; trigger point therapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinding will be used in which only the researcher doing the study knows which treatment or intervention the participant is receiving until the trial is over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Following physiotherapy will be given to the participants in this group for 6 weeks, 2 times a week:
  1. Positional Release Technique 2. Ultrasound 3. Cold Packs 4. Hip Strengthening Exercises 5. Knee Strengthening exercises
  Interventions: Other: Physiotherapy
- Comparator (Active Comparator): Following physiotherapy will be given to the participants in this group for 6 weeks, 2 times a week:
  1. Myofascial Release Technique 2. Ultrasound 3. Cold Packs 4. Hip Strengthening Exercises 5. Knee Strengthening exercises
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Treatment will be given in 3 sessions per week for 6 weeks with home exercise program and participants will be provided with exercises sheets to remember the exercises.
  The selected outcome measure will be taken on baseline (initial visit) and 6th week (post intervention)

SUMMARY:
Patellofemoral pain syndrome is a condition of misleading diagnosis. It mostly affects individuals with ages between 18-40 years. It is believed that much work has been done on the joint itself in treating the Quadriceps muscles and triggers related to it but now literature is focusing on the segmental involvement, where weakness of the hip abductors and lateral rotators play a major role. Therefore, interventions used for treating this syndrome should include on focusing the hip muscles for trigger point therapy as well as strengthening them in increasing the stability of the hip and pelvis to reduce excessive valgus forces on the knee.

DETAILED DESCRIPTION:
Literature regarding Gluteus Medius trigger point is quite scarce especially in alleviating the pain related to Patellofemoral Pain Syndrome. The management of Patellofemoral Pain Syndrome includes a segmental treatment, giving special focus to the lateral rotators and abductors of the hip especially Gluteus Medius muscle, rather than treating the Patellofemoral Joint itself. It will help in improving the pain of the subjects suffering from this syndrome effectively, and within a shorter duration of time. It will also provide the practicing physiotherapist with an insight for treating such patients with better outcomes. Myofascial Trigger Points of the Gluteus Medius are important contributing factors in the management of Patellofemoral Pain Syndrome which is identified in a single study as per author's knowledge. But the treatment used to release the trigger point of Gluteus Medius in managing this syndrome has not yet been explored. So, this study will compare two well-known treatments in comprehending which one of the two techniques have better effects on the population to be studied. Written consent will be taken from all the study participants. Simple randomization technique will be used through "Randomization Main" software and randomization sheet will be generated. 60 participants with patellofemoral pain syndrome having Gluteus Medius trigger point will be randomly allocated in two equal group.

ELIGIBILITY:
Inclusion Criteria:

* Anterior knee pain >1month and <3 month
* Pain in activities like ascending & descending stairs, running or sports activity & prolonged sitting
* Presence of Gluteus Medius trigger point in the affected limb
* Age group 18-40 years
* Both genders

Exclusion Criteria:

* Dislocation of Patella
* Damaged cartilage and ligament of Knee Joint
* Soft tissue injury related to Knee
* Any knee or hip surgery
* Lumbar spine dysfunction
* Sacroiliac joint dysfunction
* Pelvic malalignment
* Flat foot
* Chondromalacia patellae
* Young onset Osteoarthritis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Anterior Knee pain Scale | Baseline and end of intervention (6th week)
  It is 13-item questionnaire with different categories relating various levels of individual's current knee function. Score ranges from 1 representing severe disability to 100 representing no disability.
Visual Analog Scale | Baseline and end of intervention (6th week)
  A subjective psychometric response scale used to measure discrete behavioral or physiological phenomena based on linear numerical gradient in measuring the intensity of pain.
Pain Pressure Threshold | Baseline and end of intervention (6th week)
  It is the amount of direct pressure required in eliciting a response in pain on a selected area obtained by an Algometer in kilograms (kg.)

SECONDARY OUTCOMES:
Muscle strength | Baseline and end of intervention (6th week)
  In kilograms (kg.) obtained by Hand Held Dynamometer
World Health Organization Quality of Life Questionnaire- Brief | Baseline and end of intervention (6th week)
  An integrated instrument used to evaluate health related quality of life. It is a 26-item version of the WHOQOL-100 assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Kumar, MSAPT, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Results will be explored through publications.
Supporting Information: Study Protocol, SAP
Time Frame: Results will be explored through publications.
Access Criteria: Results will be explored through publications.

REFERENCES:
- [Derived] Kumar PR, Soomro RR. Comparing the effects of positional versus myofascial release of gluteus medius to manage patellofemoral pain syndrome: single blinded randomized clinical trial. J Pak Med Assoc. 2024 Feb;74(2):216-223. doi: 10.47391/JPMA.8654. PMID 38419216